CLINICAL TRIAL: NCT05037838
Title: Strain Analysis for Assessment of Myocardic Dysfunction During Orthotopic Liver Transplantation
Acronym: STRAIN ETO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2021_002
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-06

CONDITIONS: Myocardial Dysfunction; Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient undergoing a liver transplantation: Patients undergoing a liver transplantation and able to have a transesopahageal ultrasound
  Interventions: Procedure: Longitudinal strain obtained thanks to transesophageal ultrasound data recorded during liver transplantation

INTERVENTIONS:
Procedure: Longitudinal strain obtained thanks to transesophageal ultrasound data recorded during liver transplantation — Longitudinal strain of Left Ventricule and longitudinal strain of Right Ventricule free wall obtained thanks to TransEosophagal Ultrasound performed during the Liver Transplant

SUMMARY:
Mycocardial systolic function (contractility) is an essential element of cardio-circulatory physiology during major visceral surgery, in particular during liver transplantation during which several factors are likely to be at the origin of a ventricular dysfunction: acute hemorrhage, major volume changes, acute pulmonary arterial hypertension and ischemia-reperfusion syndrome.

Ventricular dysfunction is an underestimated intraoperative liver transplantation phenomenon while it constitutes a risk factor for peroperative and postoperative morbidity and mortality established that graft function can be compromised through the phenomena of low cardiac output and hepatic congestion.

Also, better analyzing myocardial systolic function during liver transplantation could guide practitioners in the treatments to be undertaken, evaluate their effects and diagnose various complications.

In addition, the usual cardiac output measurement systems (transpulmonary thermodilution techniques and pulse wave contour analysis) are poorly suited to liver transplantation. Frequent variations in blood volume, vasomotor tone and temperature require regular recalibrations and prevent a continuous and reliable estimate of cardiac output.

Thus, the choice of hemodynamic monitoring during liver transplantation performed in our center is transesophageal ultrasound, a semi-invasive method with a favorable benefit-risk ratio in this category of the population. However, analysis of right ventricular systolic function by classical indices is difficult in transesophageal ultrasound for reasons of alignment of the ultrasound shot on the right ventricular. The analysis of left ventricular systolic function is complex due to the sudden variations in volume and the difficulty in carrying out planimetry measurements in real time.

Myocardial strain imaging has been developed in recent years and is widely validated for the assessment of left ventricular contractile function. It was subsequently applied to the exploration of the right ventricular. Its measurement can be performed from recordings on dedicated software.

Thus, the strain could make it possible to better assess myocardial systolic dysfunction in liver per-transplantation from the transesophageal echographic loops recorded in current practice at the different operating times. Strain measurements will be carried out a posteriori from the images which are acquired in a standard way during the operation.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years old and more
* Patients undergoing a liver transplantation

Exclusion Criteria:

* Contraindication to transesophageal ultrasound
* Refusal to participate
* Age <18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
variations of strain | The variations will be observed thanks to measurements done before incision, during the dissection phase, during the anhepatic period, during the reperfusion phase, during the biliary reconstruction and finally after the patient closure
  Variations of left ventricular longitudinal strain and right ventricular free wall longitudinal strain obtained with transesophageal ultrasound data during each phase of orthotopic liver transplantation, The primary endpoint is to objective a myocardial dysfunction comparatively to baseline assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital de la Croix Rousse, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared